CLINICAL TRIAL: NCT05884801
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of QLS1103 in Subjects With Advanced Solid Tumors
Brief Title: Phase I Study of QLS1103 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLS1103-101
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS1103 Dose Escalation and Expansion (Experimental)
  Interventions: Drug: QLS1103

INTERVENTIONS:
Drug: QLS1103 — Oral dose

SUMMARY:
This study is a phase I, dose escalation and dose expansion study of QLS1103, to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of QLS1103 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form;
* 2. Aged ≥18 years old;
* 3. Histologically or cytologically confirmed advanced or recurrent or metastatic solid tumor;
* 4. Failure of adequate standard treatment, or no effective standard treatment;
* 5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
* 6. Life expectancy ≥12 weeks;

Exclusion Criteria:

* 1. Subjects received systemic anticancer therapy within 4 weeks prior to the first dose;
* 2. Subjects received experimental medication or therapy within 4 weeks prior to the first dose;
* 3. Subjects received major surgery within 4 weeks prior to the first dose;
* 4. Persistent toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >1 severity that is related to prior therapy;
* 5. Cardiovascular and cerebrovascular diseases with clinical significance;
* 6. Active gastrointestinal disease or other conditions that significantly interfere with drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 21 Days (first cycle)
Recommended dose for phase II (RP2D) | Up to 24 approximately months
Adverse events(AEs) / Serious adverse events(SAEs) | Up to 24 approximately months

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of QLS1103 | Up to approximately 2 years
Time of maximum observed plasma concentration (Tmax) of QLS1103 | Up to approximately 2 years
Area under the plasma concentration-time curve (AUC) of QLS1103 | Up to approximately 2 years
Objective response rate (ORR) | Up to approximately 2 years
Disease control rate (DCR) | Up to approximately 2 years
Duration of response (DOR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China